CLINICAL TRIAL: NCT03115866
Title: FRUVEDomics Study: Use of a Behavioral Nutrition Intervention in Young Adults to Identify Modifiable Metabolomics and Microbiome Risk
Brief Title: FRUVEDomics: Behavioral Intervention in Young Adults to Identify Metabolomics and Microbiome Risk
Acronym: FRUVEDomics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Collaborators: University of Tennessee (Other); University of New Hampshire (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 1409433435; 2014-67001-21851 (Other Grant/Funding Number: USDA National Institute of Food and Agriculure)
Record Dates: First submitted 2017-04-05; First posted 2017-04-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Metabolic Syndrome
Keywords: Healthy Diet; Fruits and Vegetables; Metabolome; Microbiome; Young Adults
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: 2 interventions evaluated against the other and a control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FRUVED (Experimental): Individuals that are at risk for metS and those with metS went through an 8-week dietary intervention called FRUVEDomics to increase fruit and vegetable consumption measuring metabolome and microbiome markers with health-related behaviors. In this arm, individuals were assigned to a diet with 50% fruit and vegetables.
  Interventions: Behavioral: FRUVEDomics
- FRUVED + LRC (Experimental): Individuals at risk for metS and those with metS went through an 8-week dietary intervention called FRUVEDomics to increase fruit and vegetable consumption measuring metabolome and microbiome markers with health-related behaviors. In this arm, individuals were assigned to a diet of 50% fruit and vegetables plus low refined carbohydrates.
  Interventions: Behavioral: FRUVEDomics
- FRUVED + LF (Experimental): Individuals at risk for metS and those with metS went through an 8-week dietary intervention called FRUVEDomics to increase fruit and vegetable consumption measuring metabolome and microbiome markers with health-related behaviors. In this arm, individuals were assigned to a diet of 50% fruit and vegetables plus low fat.
  Interventions: Behavioral: FRUVEDomics

INTERVENTIONS:
Behavioral: FRUVEDomics — FRUVEDomics is a behavioral nutrition intervention in young adults 'at risk for metS' and young adults 'with metS' to identify modifiable metabolomics and microbiome risk. Group nutrition education including basic nutrition for the prescribed intervention, culinary tool kit distribution, sample budget and grocery shopping tips were delivered to each participant group prior to the start of the intervention. Participants underwent individual weekly consultations with a Registered Dietitian Nutritionist using food logs, food pictures and receipt management, to assess adherence and cost of the intervention.

SUMMARY:
Rates of obesity and the metabolic syndrome are increasing in the young adult population (years 18-28). Modifying diet, especially increasing fruit and vegetable intake, can help assist in health maintenance and disease prevention. The purpose of this project is to evaluate the impact of the FRUVEDomics behavior intervention on dietary behaviors and metabolic parameters on young adults "at-risk" of disease. FRUVEDomics is an 8-week free-living dietary intervention, based on the USDA Dietary Guidelines for Americans and driven by the Social Cognitive Theory, conducted in young adults (18-28 years old) at West Virginia University. Individuals were recruited if they had pre-existing poor nutritional habits. A metabolic syndrome risk screening score was given to participants at baseline to measure "risk" status for chronic disease. Subjects were randomized into one of three nutritional intervention groups: 1) "FRUVED" (50% fruit & vegetable), 2) "FRUVED+LRC" (50% fruit & vegetable plus low refined carbohydrate), and 3) "FRUVED+LF" (50% fruit & vegetable plus low fat). Anthropometrics, surveys, venous blood samples and body composition were collected before and after the intervention. Group nutrition education including basic nutrition for the prescribed intervention, culinary tool kit distribution, sample budget and grocery shopping tips were delivered to each participant group prior to the start of the intervention. Participants underwent individual weekly consultations with a Registered Dietitian Nutritionist using food logs, food pictures and receipt management, to assess adherence and cost of the intervention.

DETAILED DESCRIPTION:
Background: Rates of obesity and the metabolic syndrome are increasing in the young adult population (years 18-28), further creating a need for interventions that will improve later quality of life. Modifying diet, especially increasing fruit and vegetable intake, can help assist in health maintenance and disease prevention. In the past decade, there has been considerable research on behavior interventions focusing on dietary change for the promotion of health. However, successful theory-based dietary behavioral interventions for young adults who follow poor lifestyle habits, are limited. The purpose of this paper is to evaluate the impact of the FRUVEDomics pilot study on dietary behaviors and metabolic parameters on young adults "at-risk" of disease.

Methods: An 8-week free-living dietary intervention, based on the USDA Dietary Guidelines for Americans and driven by the Social Cognitive Theory, was conducted in young adults (18-28 years old) at West Virginia University. Individuals were recruited if they had pre-existing poor nutritional habits. A metabolic syndrome risk screening score was given to participants at baseline to measure "risk" status for chronic disease. Subjects (n=36) were randomized into one of three nutritional intervention groups; 1) "FRUVED" (50% fruit & vegetable), 2) "FRUVED+LRC" (50% fruit & vegetable plus low refined carbohydrate), and 3) "FRUVED+LF" (50% fruit & vegetable plus low fat). Anthropometrics, surveys, venous blood samples and body composition were collected before and after the intervention. Group nutrition education including basic nutrition for the prescribed intervention, culinary tool kit distribution, sample budget and grocery shopping tips were successfully delivered to each participant group prior to the start of the intervention. Participants underwent individual weekly consultations with a Registered Dietitian Nutritionist using food logs, food pictures and receipt management, to assess adherence and cost of the intervention.

Specific Aim: Identify novel metabolomic and microbiome phenotypes in response to fruit and vegetable diet intervention in young adults with and without metabolic syndrome (MetS).

Hypothesis 1: Diet consisting of 50% fruit & vegetable consumption (FRUVED diet) will improve metabolic health as evidenced by lower plasma concentrations of adipokines, inflammatory mediators, and ceramides.

Hypothesis 2. Diet induced changes in the metabolome and micobiome will reveal novel phenotypes that have the potential to be used as new diagnostic biomarkers to distinguish between MetS and healthy adolescents.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 28 years of age
* either showing evidence of metabolic syndrome or at risk for metabolic syndrome

Exclusion Criteria:

* no evidence of metabolic syndrome or of being at-risk for metabolic syndrome

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Change in metabolic parameters at 8 weeks | Baseline (T0), Week 3 (T1), Week 5 (T2), and Post Week 8 (T3)
  Metabolomic measures via blood sample

SECONDARY OUTCOMES:
Change in microbiome parameters at 8 weeks | Baseline (T0), Week 3 (T1), Week 5 (T2), and Post Week 8 (T3)
  Microbiome measures via stool sample
Change in Weight and BMI at 8 weeks | 8 weeks
  calculation with body weight and height
Change in Blood pressure at 8 weeks | 8 weeks
  Blood pressure, standard measurement equipment
Change in Arterial stiffness at 8 weeks | 8 weeks
  Measured via dopler

CONTACTS AND LOCATIONS:
Overall Officials: Melissa D. Olfert, DrPH, RDN, Principal Investigator — West Virginia University

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD at this time.

REFERENCES:
- [Background] Tabas I. Cholesterol in health and disease. J Clin Invest. 2002 Sep;110(5):583-90. doi: 10.1172/JCI16381. No abstract available. PMID 12208856
- [Background] Barsh GS, Schwartz MW. Genetic approaches to studying energy balance: perception and integration. Nat Rev Genet. 2002 Aug;3(8):589-600. doi: 10.1038/nrg862. No abstract available. PMID 12154382
- [Background] Seeman E. Pathogenesis of bone fragility in women and men. Lancet. 2002 May 25;359(9320):1841-50. doi: 10.1016/S0140-6736(02)08706-8. PMID 12044392
- [Background] Catalan U, Rodriguez MA, Ras MR, Macia A, Mallol R, Vinaixa M, Fernandez-Castillejo S, Valls RM, Pedret A, Griffin JL, Salek R, Correig X, Motilva MJ, Sola R. Biomarkers of food intake and metabolite differences between plasma and red blood cell matrices; a human metabolomic profile approach. Mol Biosyst. 2013 Jun;9(6):1411-22. doi: 10.1039/c3mb25554a. Epub 2013 Mar 14. PMID 23493899
- [Background] German JB, Roberts MA, Fay L, Watkins SM. Metabolomics and individual metabolic assessment: the next great challenge for nutrition. J Nutr. 2002 Sep;132(9):2486-7. doi: 10.1093/jn/132.9.2486. No abstract available. PMID 12221197
- [Background] Morrow DA. Fat cow syndrome. J Dairy Sci. 1976 Sep;59(9):1625-9. doi: 10.3168/jds.S0022-0302(76)84415-3. PMID 965540
- [Background] McCann JP, Reimers TJ. Insulin response to glucose in estrous and diestrous obese and lean heifers. J Anim Sci. 1985 Sep;61(3):619-23. doi: 10.2527/jas1985.613619x. PMID 3905736
- [Background] Despres JP, Lemieux I. Abdominal obesity and metabolic syndrome. Nature. 2006 Dec 14;444(7121):881-7. doi: 10.1038/nature05488. PMID 17167477
- [Background] Holland WL, Summers SA. Sphingolipids, insulin resistance, and metabolic disease: new insights from in vivo manipulation of sphingolipid metabolism. Endocr Rev. 2008 Jun;29(4):381-402. doi: 10.1210/er.2007-0025. Epub 2008 May 1. PMID 18451260
- [Background] Long SD, Pekala PH. Lipid mediators of insulin resistance: ceramide signalling down-regulates GLUT4 gene transcription in 3T3-L1 adipocytes. Biochem J. 1996 Oct 1;319 ( Pt 1)(Pt 1):179-84. doi: 10.1042/bj3190179. PMID 8870666
- [Background] Kanety H, Hemi R, Papa MZ, Karasik A. Sphingomyelinase and ceramide suppress insulin-induced tyrosine phosphorylation of the insulin receptor substrate-1. J Biol Chem. 1996 Apr 26;271(17):9895-7. doi: 10.1074/jbc.271.17.9895. PMID 8626623
- [Background] Shah C, Yang G, Lee I, Bielawski J, Hannun YA, Samad F. Protection from high fat diet-induced increase in ceramide in mice lacking plasminogen activator inhibitor 1. J Biol Chem. 2008 May 16;283(20):13538-48. doi: 10.1074/jbc.M709950200. Epub 2008 Mar 22. PMID 18359942
- [Background] Zhang HH, Halbleib M, Ahmad F, Manganiello VC, Greenberg AS. Tumor necrosis factor-alpha stimulates lipolysis in differentiated human adipocytes through activation of extracellular signal-related kinase and elevation of intracellular cAMP. Diabetes. 2002 Oct;51(10):2929-35. doi: 10.2337/diabetes.51.10.2929. PMID 12351429
- [Background] Laurencikiene J, van Harmelen V, Arvidsson Nordstrom E, Dicker A, Blomqvist L, Naslund E, Langin D, Arner P, Ryden M. NF-kappaB is important for TNF-alpha-induced lipolysis in human adipocytes. J Lipid Res. 2007 May;48(5):1069-77. doi: 10.1194/jlr.M600471-JLR200. Epub 2007 Feb 1. PMID 17272828
- [Background] Bocci G, Fioravanti A, Orlandi P, Di Desidero T, Natale G, Fanelli G, Viacava P, Naccarato AG, Francia G, Danesi R. Metronomic ceramide analogs inhibit angiogenesis in pancreatic cancer through up-regulation of caveolin-1 and thrombospondin-1 and down-regulation of cyclin D1. Neoplasia. 2012 Sep;14(9):833-45. doi: 10.1593/neo.12772. PMID 23019415
- [Background] Sung HK, Doh KO, Son JE, Park JG, Bae Y, Choi S, Nelson SM, Cowling R, Nagy K, Michael IP, Koh GY, Adamson SL, Pawson T, Nagy A. Adipose vascular endothelial growth factor regulates metabolic homeostasis through angiogenesis. Cell Metab. 2013 Jan 8;17(1):61-72. doi: 10.1016/j.cmet.2012.12.010. PMID 23312284
- [Background] Olfert IM, Howlett RA, Tang K, Dalton ND, Gu Y, Peterson KL, Wagner PD, Breen EC. Muscle-specific VEGF deficiency greatly reduces exercise endurance in mice. J Physiol. 2009 Apr 15;587(Pt 8):1755-67. doi: 10.1113/jphysiol.2008.164384. Epub 2009 Feb 23. PMID 19237429
- [Background] Olfert IM, Howlett RA, Wagner PD, Breen EC. Myocyte vascular endothelial growth factor is required for exercise-induced skeletal muscle angiogenesis. Am J Physiol Regul Integr Comp Physiol. 2010 Oct;299(4):R1059-67. doi: 10.1152/ajpregu.00347.2010. Epub 2010 Aug 4. PMID 20686173
- [Background] Haus JM, Kashyap SR, Kasumov T, Zhang R, Kelly KR, Defronzo RA, Kirwan JP. Plasma ceramides are elevated in obese subjects with type 2 diabetes and correlate with the severity of insulin resistance. Diabetes. 2009 Feb;58(2):337-43. doi: 10.2337/db08-1228. Epub 2008 Nov 13. PMID 19008343
- [Background] Blachnio-Zabielska AU, Pulka M, Baranowski M, Nikolajuk A, Zabielski P, Gorska M, Gorski J. Ceramide metabolism is affected by obesity and diabetes in human adipose tissue. J Cell Physiol. 2012 Feb;227(2):550-7. doi: 10.1002/jcp.22745. PMID 21437908
- [Background] Gatt S, Dagan A. Cancer and sphingolipid storage disease therapy using novel synthetic analogs of sphingolipids. Chem Phys Lipids. 2012 May;165(4):462-74. doi: 10.1016/j.chemphyslip.2012.02.006. Epub 2012 Feb 23. PMID 22387097
- [Background] Brindley DN, Lin FT, Tigyi GJ. Role of the autotaxin-lysophosphatidate axis in cancer resistance to chemotherapy and radiotherapy. Biochim Biophys Acta. 2013 Jan;1831(1):74-85. doi: 10.1016/j.bbalip.2012.08.015. Epub 2012 Aug 29. PMID 22954454
- [Background] Morrell JS, Byrd-Bredbenner C, Quick V, Olfert M, Dent A, Carey GB. Metabolic syndrome: comparison of prevalence in young adults at 3 land-grant universities. J Am Coll Health. 2014;62(1):1-9. doi: 10.1080/07448481.2013.841703. PMID 24313691
- [Background] National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). Third Report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III) final report. Circulation. 2002 Dec 17;106(25):3143-421. No abstract available. PMID 12485966
- [Background] Turconi G, Guarcello M, Berzolari FG, Carolei A, Bazzano R, Roggi C. An evaluation of a colour food photography atlas as a tool for quantifying food portion size in epidemiological dietary surveys. Eur J Clin Nutr. 2005 Aug;59(8):923-31. doi: 10.1038/sj.ejcn.1602162. PMID 15928683
- [Background] Swanson M. Digital photography as a tool to measure school cafeteria consumption. J Sch Health. 2008 Aug;78(8):432-7. doi: 10.1111/j.1746-1561.2008.00326.x. PMID 18651930
- [Background] Cockburn AF, Dehlin JM, Ngan T, Crout R, Boskovic G, Denvir J, Primerano D, Plassman BL, Wu B, Cuff CF. High throughput DNA sequencing to detect differences in the subgingival plaque microbiome in elderly subjects with and without dementia. Investig Genet. 2012 Sep 21;3(1):19. doi: 10.1186/2041-2223-3-19. PMID 22998923
- See also: Olfert Research Lab — http://melissa-olfert.davis.wvu.edu/research-projects/fruvedomics